CLINICAL TRIAL: NCT03341962
Title: A Phase 2, Multicenter, Randomized, Double-blind, Placebo-controlled, Dose-finding Study to Evaluate the Efficacy and Safety of IMU-838 for Induction and Maintenance Therapy in Moderate-to-severe Ulcerative Colitis
Brief Title: Phase 2 Dose-finding IMU-838 for Ulcerative Colitis
Acronym: CALDOSE-1
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Considering the efficacy results of the induction phase (allowed use of corticosteroids as concomitant medication) in the study population and since IMU-838 did not show superiority over placebo, the OLE was prematurely closed by the sponsor.
Sponsor: Immunic AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P2-IMU-838-UC; P2-IMU-838-UC (Other: Sponsor protocol ID); 2017-003703-22 (EudraCT Number)
Record Dates: First submitted 2017-11-08; First posted 2017-11-14 (Actual); Results first posted 2024-03-05 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-02

CONDITIONS: Ulcerative Colitis
Keywords: Ulcerative Colitis; IMU-838; vidofludimus calcium
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- 10 mg IMU-838 (Induction) (Experimental): Two 5 mg tablets once daily of IMU-838 for 10 to 22 weeks depending on symptomatic remission at Weeks 10 or 22.
  Patients will receive only half of their assigned full dose during the first week of treatment.
  Interventions: Drug: IMU-838
- 30 mg IMU-838 (Induction) (Experimental): Two 15 mg tablets once daily of IMU-838 for 10 to 22 weeks depending on symptomatic remission at Weeks 10 or 22.
  Patients will receive only half of their assigned full dose during the first week of treatment.
  Interventions: Drug: IMU-838
- 45 mg IMU-838 (Induction) (Experimental): Two 22.5 mg tablets once daily of IMU-838 for 10 to 22 weeks depending on symptomatic remission at Weeks 10 or 22.
  Patients will receive only half of their assigned full dose during the first week of treatment.
  Interventions: Drug: IMU-838
- placebo (Induction) (Placebo Comparator): The placebo tablets will be identical to the IMU-838 tablets in terms of appearance, constitution of inactive ingredients, and packaging.
  Interventions: Drug: Placebo
- 10 mg IMU-838 (Maintenance) (Experimental): Two 5 mg tablets once daily of IMU-838 until Week 50 or ulcerative colitis relapse.
  Interventions: Drug: IMU-838
- 30 mg IMU-838 (Maintenance) (Experimental): Two 15 mg tablets once daily of IMU-838 until Week 50 or ulcerative colitis relapse.
  Interventions: Drug: IMU-838
- placebo (Maintenance) (Placebo Comparator): The placebo tablets will be identical to the IMU-838 tablets in terms of appearance, constitution of inactive ingredients, and packaging. Patients who have received placebo during the induction phase will be 're-randomized' to continue to receive placebo (in a blinded fashion).
  Interventions: Drug: Placebo
- 30 mg IMU-838 (Open-label) (Experimental): Two 15 mg tablets once daily of IMU-838 or one 30 mg tablet IMU-838 once daily for up to 10 years and up to 3 years in UK sites
  Interventions: Drug: IMU-838

INTERVENTIONS:
Drug: IMU-838 — IMU-838 tablet
  Other Names: IM90838; vidofludimus calcium
  Arms: 10 mg IMU-838 (Induction); 10 mg IMU-838 (Maintenance); 30 mg IMU-838 (Induction); 30 mg IMU-838 (Maintenance); 30 mg IMU-838 (Open-label); 45 mg IMU-838 (Induction)
Drug: Placebo — Tablets manufactured to mimic IMU-838 tablets
  Other Names: Placebo (for IMU-838)
  Arms: placebo (Induction); placebo (Maintenance)

SUMMARY:
This is a phase 2, multicenter, randomized, double-blind, placebo-controlled, dose-finding study to evaluate the efficacy and safety of IMU-838 for induction and maintenance therapy with an option for open-label treatment extension in moderate-to-severe ulcerative colitis (CALDOSE-1).

DETAILED DESCRIPTION:
The investigational medicinal product (IMP) IMU-838 (vidofludimus calcium) is a new compound that selectively inhibits the human enzyme dihydroorotate dehydrogenase (DHODH). Dihydroorotate dehydrogenase plays a major role in the de-novo pyrimidine synthesis and is specifically expressed at high levels in proliferating or activated lymphocytes. Resting lymphocytes satisfy their pyrimidine requirements through a DHODH-independent salvage pathway. Thus, IMU-838-mediated DHODH inhibition selectively affects activated, rapidly proliferating lymphocytes. The metabolic stress secondary to DHODH inhibition leads to a reduction of pro-inflammatory cytokine release including interleukin (IL)-17 (IL-17A and IL-17F) and interferon gamma (IFNγ), and to an increased apoptosis in activated lymphocytes.

This is a phase 2, multicenter, randomized, double-blind, and placebo-controlled trial in patients with moderate-to-severe UC with an option for open-label treatment extension. The study comprises a blinded induction phase to establish the optimal dose of IMU-838 to induce response and remission, a blinded maintenance phase to evaluate the potential of IMU-838 to maintain remission until Week 50, and an open-label treatment extension arm for all patients who discontinue the blinded phase as scheduled or prematurely, subject to certain restrictions. A subset of patients will undergo a pharmacokinetic (PK) period at the start of the open-label period to establish a full single-dose PK profile.

ELIGIBILITY:
INCLUSION CRITERIA:

Induction phase

1. Male and female patients, aged 18 - 80 years
2. UC diagnosed more than 3 months before Screening (Day-30) as documented in the medical chart
3. Previous treatment failure defined as:

   1. Patient had an inadequate response with, lost response to, or was intolerant to approved or experimental immunomodulators (azathioprine, 6-mercaptopurine, 6-thioguanine, methotrexate, or tofacitinib) or biologics (no more than 2 treatment failures with biologic drugs i.e. anti-tumor necrosis factor α antibodies [infliximab, adalimumab, golimumab and their biosimilars], vedolizumab, or certain experimental antibodies [ustekinumab]); or
   2. Patient had an inadequate response to, was intolerant to, or is corticosteroid dependent (corticosteroid-dependent patients are defined as i) unable to reduce steroids below the equivalent of prednisolone 10 mg/day within 3 months of starting steroids, without recurrent active disease, or ii) who have a relapse within 3 months of stopping steroids.)
4. Active disease defined as

   a. Mayo stool frequency score of ≥2 at Screening Visit 1 b. Mayo rectal bleeding score of ≥1 at Screening Visit 1 c. modified Mayo endoscopy subscore of ≥2 at the screening flexible sigmoidoscopy (endoscopy assessed by an independent central reader blinded to screening center and patient information)
5. Endoscopic appearance typical for UC and extending >15 cm from the anal verge as confirmed by an independent central reader (blinded to screening center and patient information)
6. Laboratory values: Neutrophil count >1500 cells/µL, platelet count ≥100 000 /mm3, serum creatinine <1.5 x upper limit of normal (ULN), total bilirubin, alanine aminotransferase (ALT), and gamma-glutamyl transferase (GGT) <1.5 x ULN
7. Female patients must:

   a. Be of non-child-bearing potential i.e. surgically sterilized (hysterectomy, bilateral salpingectomy, bilateral oophorectomy at least 6 weeks before Screening) or post-menopausal (where postmenopausal is defined as no menses for 12 months without an alternative medical cause), or

   b. If of child-bearing potential, must have a negative pregnancy test at Screening (blood test) and before the first study drug administration (Day 0 urine test). They must agree not to attempt to become pregnant, must not donate ova, and must use a highly effective contraceptive method 2 months before Screening, during treatment with IMU-838, and at least 3 months after the last dose of study therapy

   Highly effective forms of birth control are those with a failure rate less than 1% per year and include:

   - oral, intravaginal, or transdermal combined (estrogen and progestogen containing) hormonal contraceptives associated with inhibition of ovulation
   * oral, injectable, or implantable progestogen-only hormonal contraceptives associated with inhibition of ovulation
   * intrauterine device or intrauterine hormone-releasing system
   * bilateral tubal occlusion
   * vasectomized partner (i.e. the patient's male partner has undergone effective surgical sterilization before the female patient entered the clinical trial and he is the sole sexual partner of the female patient during the clinical trial)
   * sexual abstinence (acceptable only if it is the patient's usual form of birth control/lifestyle choice) 8. Male patients must agree not to father a child or to donate sperm starting at Screening and throughout the clinical trial and for 3 months after the last dose of study medication.
8. Male patients must also either

   - abstain from sexual intercourse with a female partner (acceptable only if it is the patient's usual form of birth control/lifestyle choice), or

   - use adequate barrier contraception during treatment with IMU-383 and for at least 3 months after the last dose of study medication

   For Poland and the UK the following additional requirement apply:
   * if male patients have a female partner of childbearing potential, the partner should use a highly effective contraceptive method as outlined in inclusion criterion 7

   And additionally, for Poland only:
   * if male patients have a pregnant partner, they must use condoms while taking study medication to avoid exposure of the fetus to study medication
9. Ability to understand and comply with study procedures and restrictions
10. The patient is legally competent, has been informed of the nature, the scope and the relevance of the study, voluntarily agrees to participation and the study's provisions and has duly signed the informed consent form

Maintenance phase

1. Symptomatic remission achieved at Week 10 or Week 22 of the induction phase

Open-label treatment extension arm

1. Patient is in the induction phase, had received at least 6 weeks of blinded study treatment and completed the sigmoidoscopy (incl. biopsy) regularly scheduled at Week 10/End of Induction, and has neither reached symptomatic remission nor symptomatic response

OR

Patient is in the extended induction phase, had completed all Week 10 assessments, and has not reached symptomatic remission during or at the end of the extended induction phase, Or Patient is in the maintenance phase and discontinues from the maintenance phase due to symptomatic UC relapse or other reasons with a flexible sigmoidoscopy performed at discontinuation (if the previous sigmoidoscopy had been performed more than 4 weeks before discontinuation)

OR

Patient has completed the maintenance phase as scheduled (including all Week 50 assessments)

EXCLUSION CRITERIA:

Gastrointestinal exclusion criteria

1. Diagnosis of Crohn's disease, inflammatory bowel disease type unclassified, ischemic colitis, microscopic colitis, radiation colitis or diverticular disease-associated colitis
2. Ileostomy, colostomy, or known fixed symptomatic stenosis of the intestine
3. History of colectomy with ileorectal anastomosis or ileal-pouch anal anastomosis or imminent need for colectomy (i.e. colectomy is being planned)
4. Active therapeutically uncontrollable abscess or toxic megacolon
5. Malabsorption or short bowel syndrome
6. History of colorectal cancer or colorectal dysplasia (with the exception of dysplasia in polyps which have been removed)

   Infectious disease exclusion criteria
7. Clostridium difficile (C. difficile) infection

   * Evidence of, or treatment for C. difficile infection within 30 days before first randomization
   * Positive C. difficile toxin B stool assay during the screening period
8. Treatment for intestinal pathogens other than C. difficile within 30 days prior to first randomization
9. Other chronic systemic infections

   * History of chronic systemic infections including but not limited to tuberculosis, human immunodeficiency virus (HIV), hepatitis B or C, within 6 months before Screening
   * Positive interferon-gamma release assay (IGRAs) for Mycobacterium tuberculosis at Screening
   * Positive HBsAg (hepatitis B virus surface antigen), HBcAb (hepatitis B core antibody), positive hepatitis C virus and/or HIV-antigen-antibody (HIV-Ag/Ab) test at Screening
10. Any live vaccinations within 30 days prior to study drug administration except for the influenza vaccine

    Other medical history and concomitant disease exclusion criteria
11. Known history of nephrolithiasis or underlying condition with a strong association of nephrolithiasis, including hereditary hyperoxaluria or hereditary hyperuricemia
12. Diagnosis or suspected liver function impairment which may cause, as assessed by the investigator, a potential for fluctuating liver function tests during this trial
13. Renal impairment i.e. estimated glomerular filtration rate (eGFR) ≤60 mL/min/1.73m²
14. Serum uric acid levels at Screening >1.2 x ULN (for women >6.8 mg/dL, for men >8.4 mg/dL)
15. History or clinical diagnosis of gout
16. Known or suspected Gilbert syndrome
17. Indirect (unconjugated) bilirubin ≥1.2 x ULN at Screening (i.e. ≥ 1.1 mg/dL)
18. Concurrent malignancy or prior malignancy within the previous 10 years except for the following: adequately-treated non-melanoma skin cancer and adequately-treated cervical cancer

    Therapy exclusion criteria
19. Use of any investigational product within 8 weeks or 5 x the respective half-life before first randomization, whatever is longer
20. Use of the following medications within 2 weeks before first randomization:

    1. Tofacitinib
    2. Methotrexate
    3. Mycophenolate mofetil
    4. Any calcineurin inhibitors (e.g. tacrolimus, cyclosporine, or pimecrolimus)
    5. Oral systemic corticosteroids >20 mg/day prednisolone equivalent including beclomethasone dipropionate (at >5 mg/day) and budesonide (multi-matrix [MMX] at >9 mg/day)
    6. Oral aminosalicylates (e.g. mesalazines) >4 g/day
21. Use of the following medications within 4 weeks before first randomization:

    1. Use of intravenous corticosteroids
    2. Use of thiopurines including azathioprine, mercaptopurine and 6-thioguanine
    3. Use of any rectal and topical aminosalicylates and/or budesonide
22. Use of oral systemic corticosteroids ≤20 mg/day prednisolone equivalent including beclomethasone dipropionate (at ≤5 mg/day) and budesonide (MMX at ≤9 mg/day) unless they have been used for at least 4 weeks before first randomization and at a stable dose for at least 2 weeks before first randomization
23. Oral aminosalicylates (e.g. mesalazines) ≤4 g/day unless they have been used for at least 6 weeks and with a stable dose for at least 3 weeks before first randomization
24. Use of biologics as follows:

    1. anti-tumor necrosis factor α antibodies (infliximab, adalimumab, golimumab, including their biosimilars) within 4 weeks before first randomization
    2. vedolizumab and ustekinumab within 8 weeks before first randomization
25. Use of the DHODH inhibitors leflunomide or teriflunomide within 6 months before first randomization
26. Any use of natalizumab (Tysabri™) within 12 months before first randomization
27. Use of the following concomitant medications is prohibited at Screening and throughout the duration of the trial:

    * any medication known to significantly increase urinary elimination of uric acid, in particular lesinurad (Zurampic™) as well as uricosuric drugs such as probenecid
    * treatments for any malignancy, in particular irinotecan, paclitaxel, tretinoin, bosutinib, sorafenib, enasidenib, erlotinib, regorafenib, pazopanib and nilotinib
    * any drug significantly restricting water diuresis, in particular vasopressin and vasopressin analogs
    * Rosuvastatin at doses ˃10 mg/day

    General exclusion criteria
28. History of, or current serious, severe, or unstable (acute or progressive) physical or mental illness, or any medical condition, including laboratory anomalies or renal or hepatic impairment, that may require treatment or would put the patient in jeopardy if he/she was to participate in the study
29. Known hypersensitivity to DHODH inhibitors (teriflunomide, leflunomide) or any ingredient of the investigational product
30. Pregnancy or breastfeeding
31. History of drug or alcohol abuse during the past year
32. Concurrent participation in any other clinical trial using an investigational medicinal product or medical device
33. An employee of an investigator or sponsor or an immediate relative of an investigator

Exclusion criteria for open-label treatment extension arm

1. Any ongoing, clinically significant treatment-emergent (started during the IMU-838 treatment in the blinded treatment arms) adverse event (AE) or laboratory abnormality (including blood chemistry and urinalysis) as assessed by the investigator *
2. Significant treatment or study non-compliance during induction and/or maintenance phase (as assessed by the investigator), and/or inability or unwillingness to follow instructions by study personnel as assessed by the investigator
3. Significant protocol deviations during induction and/or maintenance phase that are assessed by the investigator to negatively affect further patient cooperation in this study

   * If treatment-emergent AEs are the reason for exclusion from the open-label extension arm, the eligibility can be re-assessed up to 30 days following the last treatment in the blinded treatment arms.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 263 (Actual)
Dates: Start 2018-03-15 (Actual); Primary Completion 2022-11-16 (Actual); Study Completion 2022-11-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Muehler, Study Director — Immunic Therapeutics
Locations (131):
- United States (15):
  - Del Sol Research Management, LLC, Tucson, Arizona
  - Axis Clinical Trials, Los Angeles, California
  - Ventura Clinical Trials, Ventura, California
  - Alliance Medical Research, LLC, Lighthouse PT, Florida
  - Medley Research Associates, Medley, Florida
  - Global Life Research LLC, Miami, Florida
  - Family Clinical Trials, Pembroke Pines, Florida
  - Clinical Research Trials of Florida, Inc., Tampa, Florida
  - Atlanta Gastroenterology Associates, LLC, Atlanta, Georgia
  - McFarland Clinic, P.C., Ames, Iowa
  - Commonwealth Clinical Studies, Brockton, Massachusetts
  - PMG Research of Salisbury, LLC, Salisbury, North Carolina
  - Clinical Trials of South Carolina, Charleston, South Carolina
  - First Street Surgical Hospital, Bellaire, Texas
  - Digestive Health Specialists, Tacoma, Washington
- Albania (3):
  - Durres Regional Hospital, Durrës
  - Regional Hospital of Shkoder, Shkodër
  - University Hospital Center Mother Teresa, Tirana
- Belarus (3):
  - Gomel Regional Clinical Hospital, Homyel
  - Republican Scientific and Practical Center for Radiation Medicine and Human Ecology, Homyel
  - Vitiebsk State Order of Peoples' Friendship Medical University, Vitebsk
- Bosnia and Herzegovina (2):
  - University Clinical Centre of the Republic of Srpska, Internal Medicine Clinic, Department of Gastroenterology and Hepatology, Banja Luka
  - University Clinical Hospital Mostar, Internal Medicine Clinic, Department of Gastroenterology, Mostar
- Bulgaria (8):
  - Multiprofile Hospital for Active Treatment Blagoevgrad AD, Blagoevgrad
  - Mhat Byala, Byala
  - Multiprofile Hospital for Active Treatment "Dr. Hristo Stambolski" EOOD, Kazanlak
  - Medical Center "Medconsult Pleven" OOD, Pleven
  - Medical Center Exacta Medica, Pleven
  - University Multiprofile Hospital for Active Treatment "Sveti Georgi" EAD, Plovdiv, Gastroenterology clinic, Plovdiv
  - Medical Center "Hera" EOOD, Sofia
  - Diagnostic-Consulting Center "Convex" EOOD, Sofia
- Croatia (9):
  - General Hospital Bjelovar, Bjelovar
  - Clinical Hospital Center Osijek, Osijek
  - Clinical Hospital Center Rijeka, Rijeka
  - Clinical Hospital Center Split, Split
  - General Hospital Vukovar, Vukovar
  - Clinical Hospital Center Zagreb, Zagreb
  - Clinical Hospital Dubrava, Zagreb
  - Polyclinic Solmed Zagreb, Zagreb
  - Clinical Hospital Center Split, Zagreb
- Czechia (7):
  - Asclepiades - Interna a gastroenterologie s.r.o. - Havířov, Havířov
  - Hepato-Gastroenterologie HK, s.r.o. Poliklinika III, Hradec Králové
  - Artroscan s.r.o., Ostrava - Třebovice
  - FaraCol s.r.o. - Prague, Prague
  - MEDICON a.s. - Poliklinika Budějovická Gastroenterologie, Prague
  - Klinika ResTrial, Prague
  - Všeobecná fakultní nemocnice v Praze IV. interní klinika VFN a 1. LF UK, Prague
- Georgia (2):
  - Academician Z.Tskhakaia West Georgia National Center of Interventional Medicine, Kutaisi
  - LTD Unimedi Kakheti - Caraps Medline, Tbilisi
- Netherlands (3):
  - Amsterdam UMC, locatie AMC, Amsterdam
  - Albert Schweitzer Hospital, Dordrecht
  - Elisabeth-TweeSteden Hospital, Tilburg
- North Macedonia (2):
  - City General Hospita 8th September, Skopje
  - University Clinic for Hematology - Skopje - Macedonian Hematology Association, Skopje
- Poland (18):
  - Centrum Usług Medycznych MaxMed, Bochnia
  - Centrum Medyczne Pratia Gdynia, Gdynia
  - Centrum Medyczne Endo-med Sp. z o.o., Karczew
  - Vita Longa Sp. z o.o., Katowice
  - GLOBE Badania Kliniczne Sp. z o.o., Kłodzko
  - Salve Medica Sp. z o.o. Spółka Komandytowa, Lodz
  - Samodzielny Publiczny Szpital Kliniczny Nr 4 w Lublinie Oddział Gastroenterologii, Lublin
  - Zakład leczniczy ALLMEDICA BADANIA KLINICZNE Sp. z o.o. Sp. K., Nowy Targ
  - Etyka Ośrodek Badań Klinicznych, Olsztyn
  - Ars Medical - Szpital, Ars Medical - Ambulatorium, Piła
  - SOLUMED Centrum Medyczne, Poznan
  - Niepubliczny Zakład Opieki Zdrowotnej Centrum Medyczne HCP - Lecznictwo Stacjonarne, Poznan
  - Endoskopia Sp. z o.o., Sopot
  - Klinika Medifem, Warsaw
  - Centrum Badawcze Współczesnej Terapii, Prywatny Gabinet Lekarski dr Anna Bochenek-Mularczyk, Warsaw
  - Przychodnia Vistamed, Wroclaw
  - Centrum Medyczne OMNI Clinic Sp. z o.o. Spółka Komandytowa, Wroclaw
  - Centrum Medyczne Med-Gastr Sp. z o.o. Spółka Komandytowa, Łódz
- Portugal (3):
  - Centro Hospitalar e Universitário de Coimbra, EPE - Hospitais da Universidade de Coimbra, Coimbra
  - Hospital da Senhora da Oliveira - Guimarães, EPE, Guimarães
  - Centro Hospitalar de Entre o Douro e Vouga, EPE - Hospital São Sebastião, Santa Maria da Feira
- Romania (4):
  - S.C. MEDLIFE S.A., Sectia Gastroenterologie, Bucharest
  - Spitalul Clinic Colentina, Sectia Gastroenterologie, Bucharest
  - Institutul Clinic Fundeni, Sectia Clinica Gastroenterologie III, Bucharest
  - S.C. Cabinet Particular Policlinic Algomed SRL, Specialitatea Gastroenterologie, Timișoara
- Russia (14):
  - Kazan State Medical University, Kazan'
  - SEI HPE "Kuban State Medical University" of MoH and SD, CBHS Regional Clinical Hospital No.2, Krasnodar
  - Central Clinical Hospital of the Russian Academy of Sciences, Moscow
  - Federal Medical Biophysical Center n.a. Burnazyan, Moscow
  - Clinical Research Institution of Moscow Region named after M. F. Vladimirsky, Moscow
  - Novosibirskiy Gastrocenter, LLC, Novosibirsk
  - FSBEI HE "Military Medical Academy n.a. S.M. Kirov" under the Ministry of Defence of Russian Federation, Saint Petersburg
  - Hospital of Saint Martyr Elizaveta, Saint Petersburg
  - Research Center Eco-Safety, LLC, Saint Petersburg
  - Gastroenterological Center "Expert" LLC, Saint Petersburg
  - Saint Petersburg State Medical University named after I.P. Pavlov, Saint Petersburg
  - City Hospital No. 5 - Sochi, Sochi
  - Siberian State Medical University, Tomsk
  - Regional State Autonomous Healthcare Institution "Tomsk Regional Clinical Hospital", Tomsk
- Serbia (7):
  - Clinic for gastroenterohepatology, Belgrade
  - Clinical Hospital Center Zemun, Belgrade
  - University Hospital Center Bezaniska Kosa, Belgrade
  - Clinical Center Kragujevac, Kragujevac
  - General Hospital Leskovac, Leskovac
  - Clinical Center Nis, Niš
  - General Hospital Djordje Joanovic, Internal Deases Department, Gastroenterology, Zrenjanin
- Hospital Juan Ramón Jimenez, Huelva, Spain
- Turkey (Türkiye) (3):
  - Bezmiâlem Vakıf Üniversitesi, Fatih
  - Istanbul Universitesi Istanbul Tip Fakultesi Gastroenteroloji Bilim Dali, Fatih
  - Karadeniz Teknik Üniversitesi Tip Fakultesi, Trabzon
- Ukraine (20):
  - Public Enterprise "Dnipropetrovsk regional clinical hospital named after I.I. Mechnikova", Department of Gastroenterology (Hepatology), Dnipro
  - MNPE "Regional Clinical Hospital of Ivano-Frankivsk Regional Council", Gastroenterology Department, SHEI "Ivano-Frankivsk National Medical University", Chair of Internal Medicine #1, Ivano-Frankivsk
  - Ivano-Frankivsk City Clinical Hospital No. 1, Ivano-Frankivsk
  - Municipal Non-profit Enterprise "City Clinical Hospital #2 named after prof. O.O. Shalimova", of Kharkiv City Council, Proctology Department, Kharkiv
  - Municipal Non-profit Enterprise of Kharkiv Regional Council "Regional Clinical Hospital", Gastroenterology Department, Kharkiv
  - Private Enterprise Private Manufacturing Firm "Acinus", Treatment and diagnostic Centre, Kropyvnytskyi
  - Medical Center Medical Clinic Blagomed LLC, Kyiv
  - Kyiv City Clinical Hospital #18, Proctology Department, National Medical University named after O.O.Bogomolets, Chair of Surgery #1, Kyiv
  - Kyiv City Clinical Hospital #1, Therapeutics Department #2, Kyiv
  - Medical Centre of Limited Liability Company "Medical Centre "Dopomoga plus"", Kyiv
  - Shalimov's National Institute of surgery and transplantation, Kyiv
  - Medical Centre of Limited Liability Company "Medical Centre "Consilium Medical", clinico-consultation department, Kyiv
  - Kyiv Regional Clinical Hospital No 2, Kyiv
  - Volyn Regional Clinical Hospital, Lutsk
  - Municipal Non-profit Enterprise of Lviv Regional Council "Lviv Regional Clinical Hospital", proctology department, Danylo Galytsky Lviv National Medical University, Chair of Surgery #1, Lviv
  - KARDIOKOM Ltd., Mykolaiv
  - Transcarpathian Regional Clinical Hospital named after Andriy Novaka, gastroenterology department, Uzhhorod
  - Municipal Non-profit Enterprise "Vinnytsia Regional Clinical Hospital named after M.I. Pyrogova of Vinnytsia Regional Council, Regional Specialized Clinical Gastroenterological Center,, Vinnytsia
  - Municipal Non-profit Enterprise "Vinnytsia City Clinical Hospital #1, Gastroenterology Department, Vinnytsia National Medical University named after M.I.Pyrogova, Chair of Propaedeutics of Internal Medicine, Vinnytsia
  - Municipal Institution "Zaporizhzhska Regional Clinical Hospital" of Zaporizhzha Regional Council, gastroenterology department, Zaporizhzhya
- United Kingdom (7):
  - London North West University Healthcare NHS Trust (LNWH), St Mark's Hospital, R&D Department, Northwick Park Hospital, Harrow
  - Barts Health NHS Trust, of Royal London Hospital, London
  - University College London Hospitals NHS Foundation Trust, London
  - St Helens & Knowsley Teaching Hospitals NHS Trust, Whiston Hospital, Prescot
  - University Hospitals Coventry and Warwickshire NHS Trust, University Hospital, Shrewsbury
  - Shrewsbury and Telford Hospitals NHS Trust, Royal Shrewsbury Hospital, Shrewsbury
  - The Royal Wolverhampton NHS Trust, New Cross Hospital, Wolverhampton

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] D'Haens G, Stardelova KG, Sadiku E, Kizlova N, Skybalo S, Shehovtsova Y, Abramescu M, Vitt D, Kohlhof H, Muehler A. Vidofludimus Calcium in Patients With Moderate-to-Severe Ulcerative Colitis: A Randomized, Placebo-Controlled, Phase 2 Trial. Clin Transl Gastroenterol. 2025 Mar 1;16(3):e00813. doi: 10.14309/ctg.0000000000000813. PMID 39791563
- See also: European Medicines Agency (EMA). Guideline on the development of new medicinal products for the treatment of Ulcerative Colitis.[Online]. 2016. — https://www.ema.europa.eu/en/documents/scientific-guideline/draft-guideline-development-new-medicinal-products-treatment-ulcerative-colitis-revision-1_en.pdf
- See also: US Food and Drug Administration (FDA). Ulcerative Colitis: Clinical Trial Endpoints. Guidance for Industry.[Online]. 2016. — https://www.fda.gov/downloads/Drugs/GuidanceComplianceRegulatoryInformation/Guidances/UCM515143.pdf
- See also: American Urological Association. Guideline: Diagnosis, evaluation and follow up of asymptomatic mircrohematuria. (AMH) in adults.[Online]. 2012. — https://www.auanet.org/guidelines-and-quality/guidelines/microhematuria
- See also: EU. Regulation 2016/679 on the protection of natural persons with regard to the processing of personal data and on the free movement of such data, and repealing Directive 95/46/EC (General Data Protection Regulation). 2016; [Online]. — http://eur-lex.europa.eu/legal-content/EN/TXT/?uri=CELEX:32016R0679

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study had 3 phases, induction, maintenance and open-label. Patients who achieved symptomatic remission at Week 10 or 22 (extended) of induction phase (IP) could proceed to maintenance phase (MP). Patients who were treated for at least 6 weeks in the induction phase and fulfilled further eligibility criteria could proceed into the open label treatment extension phase (OLE).
Groups:
- 10 mg IMU-838 (Induction Phase): Two 5 mg tablets once daily of IMU-838 for 10 to 22 weeks depending on symptomatic remission at Weeks 10 or 22.
  Patients received only half of their assigned full dose during the first week of treatment.
- 30 mg IMU-838 (Induction Phase): Two 15 mg tablets once daily of IMU-838 for 10 to 22 weeks depending on symptomatic remission at Weeks 10 or 22.
  Patients received only half of their assigned full dose during the first week of treatment.
- 45 mg IMU-838 (Induction Phase): Two 22.5 mg tablets once daily of IMU-838 for 10 to 22 weeks depending on symptomatic remission at Weeks 10 or 22.
  Patients receivec only half of their assigned full dose during the first week of treatment.
- Placebo (Induction Phase): Two tablets once daily for 10 to 22 weeks depending on symptomatic remission at Weeks 10 or 22.
  Patients received only half of their assigned full dose during the first week of treatment.
- 10 mg IMU-838 (Maintenance Phase): Two 5 mg tablets once daily of IMU-838 for up to 40 weeks.
- 30 mg IMU-383 (Maintenance Phase): Two 15 mg tablets once daily of IMU-838 for up to 40 weeks.
- Placebo (Maintenance Phase): Two tablets once daily for up to 40 weeks.
- 30 mg IMU-838 (Open-label Phase): Two 15 mg tablets once daily of IMU-838.
Period: Induction Phase
Arm/Group | 10 mg IMU-838 (Induction Phase) | 30 mg IMU-838 (Induction Phase) | 45 mg IMU-838 (Induction Phase) | Placebo (Induction Phase) | 10 mg IMU-838 (Maintenance Phase) | 30 mg IMU-383 (Maintenance Phase) | Placebo (Maintenance Phase) | 30 mg IMU-838 (Open-label Phase)
Started | 67 | 67 | 66 | 63 | 0 | 0 | 0 | 0
Completed | 53 | 48 | 50 | 52 | 0 | 0 | 0 | 0
Not Completed | 14 | 19 | 16 | 11 | 0 | 0 | 0 | 0
Period: Maintenance Phase
Arm/Group | 10 mg IMU-838 (Induction Phase) | 30 mg IMU-838 (Induction Phase) | 45 mg IMU-838 (Induction Phase) | Placebo (Induction Phase) | 10 mg IMU-838 (Maintenance Phase) | 30 mg IMU-383 (Maintenance Phase) | Placebo (Maintenance Phase) | 30 mg IMU-838 (Open-label Phase)
Started (At end of the IP, 86 IMU-838 treated patients met eligibility criteria for the MP and and were re-randomized to 10 or 30 mg and 27 were "re-randomized" to the placebo group. One patient was re-randomized in the MP, but switched to the OLE before any treatment.) | 0 | 0 | 0 | 0 | 45 | 40 | 27 | 0
Completed | 0 | 0 | 0 | 0 | 35 | 29 | 21 | 0
Not Completed | 0 | 0 | 0 | 0 | 10 | 11 | 6 | 0
Period: Open-label Phase
Arm/Group | 10 mg IMU-838 (Induction Phase) | 30 mg IMU-838 (Induction Phase) | 45 mg IMU-838 (Induction Phase) | Placebo (Induction Phase) | 10 mg IMU-838 (Maintenance Phase) | 30 mg IMU-383 (Maintenance Phase) | Placebo (Maintenance Phase) | 30 mg IMU-838 (Open-label Phase)
Started (One patient was re-randomized in the MP, but switched to the OLE before any treatment. 114 patients transitioned directly from the induction phase to the OLE and received 30 mg IMU-838 and an additional 75 patients entered the OLE after the MP, resulting in a total of 190 patients in the OLE.) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 190
Completed (The study was terminated by the sponsor, therefore no patients completed the OLE.) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 190

BASELINE CHARACTERISTICS:
Population: In the IP, one patient received erroneously 30 mg IMU-838 instead of placebo and was included in the 30 mg IMU-838 group for the safety analysis set (SAF), as in participant flow, but in the placebo group for the full analysis set (FAS). Demographics and baseline characteristics were analyzed for the FAS.
  Not all participants who completed or discontinued the IP continued to the MP or OLE. Patients were re-randomized at the start of MP (except the placebo group).
Groups:
- 10 mg IMU-838 (Induction Phase): Two 5 mg tablets once daily of IMU-838 for 10 to 22 weeks.
- 30 mg IMU-838 (Induction Phase): Two 15 mg tablets once daily of IMU-838 for 10 to 22 weeks.
- 45 mg IMU-838 (Induction Phase): Two 22.5 mg tablets once daily of IMU-838 for 10 to 22 weeks.
- Placebo (Induction Phase): Two tablets once daily for 10 to 22 weeks.
- 10 mg IMU-838 (Maintenance Phase: Two 5 mg tablets once daily of IMU-838 for up to 50 weeks.
- 30 mg IMU-838 (Maintenance Phase): Two 15 mg tablets once daily of IMU-838 for up to 50 weeks.
- Placebo (Maintenance Phase): Two tablets once daily for up to 50 weeks.
- Total: Total of all reporting groups
Arm/Group | 10 mg IMU-838 (Induction Phase) | 30 mg IMU-838 (Induction Phase) | 45 mg IMU-838 (Induction Phase) | Placebo (Induction Phase) | 10 mg IMU-838 (Maintenance Phase | 30 mg IMU-838 (Maintenance Phase) | Placebo (Maintenance Phase) | 30 mg IMU-838 (Open-label Phase) | Total
Number analyzed (Participants) | 67 | 66 | 66 | 64 | 45 | 40 | 27 | 190 | 565
Age, Continuous [Median (Full Range); unit: years] — Population: FAS
  years
    Induction Phase: number analyzed (Participants) | 67 | 66 | 66 | 64 | 0 | 0 | 0 | 0 | 263
    Induction Phase | 40.0 [19 to 73] | 41.0 [21 to 77] | 40.5 [21 to 76] | 38.5 [18 to 73] |  |  |  |  | 40.0 [18 to 77]
    Maintenance phase: number analyzed (Participants) | 0 | 0 | 0 | 0 | 45 | 40 | 27 | 0 | 112
    Maintenance phase |  |  |  |  | 37.0 [19 to 76] | 39.5 [22 to 77] | 38.0 [20 to 73] |  | 38.0 [19 to 77]
    Open-label phase: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 190 | 190
    Open-label phase |  |  |  |  |  |  |  | 39.5 [18 to 77] | 39.5 [18 to 77]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: FAS
  Participants
    Induction phase: number analyzed (Participants) | 67 | 66 | 66 | 64 | 0 | 0 | 0 | 0 | 263
    Induction phase: Female | 32 | 26 | 26 | 31 |  |  |  |  | 115
    Induction phase: Male | 35 | 40 | 40 | 33 |  |  |  |  | 148
    Maintenance phase: number analyzed (Participants) | 0 | 0 | 0 | 0 | 45 | 40 | 27 | 0 | 112
    Maintenance phase: Female |  |  |  |  | 15 | 25 | 9 |  | 49
    Maintenance phase: Male |  |  |  |  | 30 | 15 | 18 |  | 63
    Open-label phase: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 190 | 190
    Open-label phase: Female |  |  |  |  |  |  |  | 83 | 83
    Open-label phase: Male |  |  |  |  |  |  |  | 107 | 107
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: FAS
  Participants
    Induction phase: number analyzed (Participants) | 67 | 66 | 66 | 64 | 0 | 0 | 0 | 0 | 263
    Induction phase: Hispanic or Latino | 0 | 1 | 0 | 3 |  |  |  |  | 4
    Induction phase: Not Hispanic or Latino | 67 | 65 | 66 | 61 |  |  |  |  | 259
    Induction phase: Unknown or Not Reported | 0 | 0 | 0 | 0 |  |  |  |  | 0
    Maintenance phase: number analyzed (Participants) | 0 | 0 | 0 | 0 | 45 | 40 | 27 | 0 | 112
    Maintenance phase: Hispanic or Latino |  |  |  |  | 0 | 0 | 0 |  | 0
    Maintenance phase: Not Hispanic or Latino |  |  |  |  | 45 | 40 | 27 |  | 112
    Maintenance phase: Unknown or Not Reported |  |  |  |  | 0 | 0 | 0 |  | 0
    Open-label phase: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 190 | 190
    Open-label phase: Hispanic or Latino |  |  |  |  |  |  |  | 3 | 3
    Open-label phase: Not Hispanic or Latino |  |  |  |  |  |  |  | 187 | 187
    Open-label phase: Unknown or Not Reported |  |  |  |  |  |  |  | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: FAS
  Participants
    Induction phase: number analyzed (Participants) | 67 | 66 | 66 | 64 | 0 | 0 | 0 | 0 | 263
    Induction phase: American Indian or Alaska Native | 0 | 0 | 0 | 0 |  |  |  |  | 0
    Induction phase: Asian | 1 | 0 | 1 | 0 |  |  |  |  | 2
    Induction phase: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 |  |  |  |  | 0
    Induction phase: Black or African American | 2 | 0 | 0 | 0 |  |  |  |  | 2
    Induction phase: White | 64 | 66 | 64 | 64 |  |  |  |  | 258
    Induction phase: More than one race | 0 | 0 | 1 | 0 |  |  |  |  | 1
    Induction phase: Unknown or Not Reported | 0 | 0 | 0 | 0 |  |  |  |  | 0
    Maintenance phase: number analyzed (Participants) | 0 | 0 | 0 | 0 | 45 | 40 | 27 | 0 | 112
    Maintenance phase: American Indian or Alaska Native |  |  |  |  | 0 | 0 | 0 |  | 0
    Maintenance phase: Asian |  |  |  |  | 0 | 0 | 0 |  | 0
    Maintenance phase: Native Hawaiian or Other Pacific Islander |  |  |  |  | 0 | 0 | 0 |  | 0
    Maintenance phase: Black or African American |  |  |  |  | 0 | 0 | 0 |  | 0
    Maintenance phase: White |  |  |  |  | 45 | 40 | 27 |  | 112
    Maintenance phase: More than one race |  |  |  |  | 0 | 0 | 0 |  | 0
    Maintenance phase: Unknown or Not Reported |  |  |  |  | 0 | 0 | 0 |  | 0
    Open-label phase: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 190 | 190
    Open-label phase: American Indian or Alaska Native |  |  |  |  |  |  |  | 0 | 0
    Open-label phase: Asian |  |  |  |  |  |  |  | 1 | 1
    Open-label phase: Native Hawaiian or Other Pacific Islander |  |  |  |  |  |  |  | 0 | 0
    Open-label phase: Black or African American |  |  |  |  |  |  |  | 1 | 1
    Open-label phase: White |  |  |  |  |  |  |  | 187 | 187
    Open-label phase: More than one race |  |  |  |  |  |  |  | 1 | 1
    Open-label phase: Unknown or Not Reported |  |  |  |  |  |  |  | 0 | 0
Region of Enrollment [Number; unit: participants] — The totals are not based on 565 participants but on the 263 participants in the induction phase. Participants in the different study phases are not exclusive.
  participants
    Romania | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
    United States | 5 | 3 | 1 | 3 | 0 | 0 | 0 | 8 | 12
    Czechia | 4 | 1 | 3 | 1 | 0 | 1 | 1 | 9 | 9
    Ukraine | 21 | 21 | 18 | 25 | 20 | 14 | 14 | 66 | 85
    United Kingdom | 4 | 2 | 0 | 4 | 1 | 0 | 2 | 9 | 10
    Belarus | 3 | 1 | 2 | 0 | 2 | 2 | 0 | 4 | 6
    Portugal | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 2
    Albania | 3 | 2 | 3 | 5 | 0 | 4 | 3 | 2 | 13
    Russia | 3 | 5 | 10 | 8 | 4 | 4 | 1 | 20 | 26
    Spain | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
    Netherlands | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 2 | 4
    North Macedonia | 5 | 2 | 2 | 1 | 1 | 1 | 0 | 6 | 10
    Poland | 11 | 20 | 12 | 12 | 9 | 9 | 4 | 42 | 55
    Bulgaria | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 3 | 3
    Serbia | 5 | 4 | 5 | 2 | 4 | 4 | 0 | 11 | 16
    Bosnia and Herzegovina | 1 | 2 | 2 | 0 | 4 | 1 | 0 | 3 | 5
    Croatia | 0 | 2 | 3 | 0 | 0 | 0 | 0 | 4 | 5
Duration of disease [Mean (Standard Deviation); unit: years] — Population: FAS, Duration of disease was only reported at Induction phase Baseline.
  years
    number analyzed (Participants) | 67 | 66 | 66 | 64 | 0 | 0 | 0 | 0 | 263
    (all) | 7.5 (7.6) | 5.8 (5.4) | 7.1 (7.4) | 5.2 (4.6) |  |  |  |  | 6.4 (6.4)
Current tobacco users [Count of Participants; unit: Participants] — Population: FAS
  Participants
    Induction phase: number analyzed (Participants) | 67 | 66 | 66 | 64 | 0 | 0 | 0 | 0 | 263
    Induction phase | 2 | 5 | 2 | 4 |  |  |  |  | 13
    Maintenance phase: number analyzed (Participants) | 0 | 0 | 0 | 0 | 45 | 40 | 27 | 0 | 112
    Maintenance phase |  |  |  |  | 1 | 0 | 0 |  | 1
    Open-label phase: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 190 | 190
    Open-label phase |  |  |  |  |  |  |  | 10 | 10
Mayo PRO-2 Score at Basline [Mean (Standard Deviation); unit: units on a scale] — The full Mayo score is composed of 4 categories (rectal bleeding, stool frequency, physician assessment, and endoscopic appearance). The Mayo patient-reported outcome (PRO) score, includes only the PROs ie, stool frequency and rectal bleeding score each rated from 0 to 3, that are added up to give a total score that ranges from 0 to 6. A higher score indicates a worse outcome. Population: FAS
  units on a scale
    Induction phase: number analyzed (Participants) | 67 | 65 | 66 | 64 | 0 | 0 | 0 | 0 | 262
    Induction phase | 4.1 (1.2) | 4.3 (1.0) | 4.3 (1.0) | 4.3 (0.9) |  |  |  |  | 4.2 (1.0)
    Maintenance phase: number analyzed (Participants) | 0 | 0 | 0 | 0 | 45 | 40 | 27 | 0 | 112
    Maintenance phase |  |  |  |  | 0.8 (0.5) | 0.9 (0.8) | 0.7 (0.5) |  | 0.8 (0.6)
    Open-label phase (Entry in open label after induction phase): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 115 | 115
    Open-label phase (Entry in open label after induction phase) |  |  |  |  |  |  |  | 3.9 (1.2) | 3.9 (1.2)
    Open-label phase (Entry in open label after maintenance phase): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 75 | 75
    Open-label phase (Entry in open label after maintenance phase) |  |  |  |  |  |  |  | 1.6 (1.7) | 1.6 (1.7)

OUTCOME MEASURES:

1. Primary Outcome: Induction Phase: Symptomatic Remission and Endoscopic Healing at Week 10
Description: Composite endpoint: Proportion of patients with both, symptomatic remission (Mayo rectal bleeding subscore = 0, and Mayo stool frequency subscore of 0 or 1) and endoscopic healing (Modified Mayo endoscopy subscore of 0 or 1) at Week 10.
  All patients who were randomized to 30 mg/day and 45 mg/day were used for the assessment of the primary efficacy endpoint
Time Frame: 10 weeks
Population: FAS
Measure: Count of Participants; unit: Participants
Groups:
- Combined IMU-838 (30 or 45 mg IMU-838, Induction Phase): Two 15 or 22.5 mg tablets once daily of IMU-838 for 10 to 22 weeks.
Arm/Group | Combined IMU-838 (30 or 45 mg IMU-838, Induction Phase) | Placebo (Induction Phase)
Number analyzed (Participants) | 116 | 57
Participants | 16 | 8
Statistical Analysis 1: Comparison: Combined IMU-838 (30 or 45 mg IMU-838, Induction Phase) vs Placebo (Induction Phase); Test type: Superiority; p = 0.5836, Cochran-Mantel-Haenszel; 1-sided exact test adjusted for stratification factors (prior use of any biologics and concurrent use of corticosteroids), α=0.097; Odds Ratio (OR) = 1.0188

2. Secondary Outcome: Induction Phase: Symptomatic Remission and Endoscopic Healing at Different Doses at Week 10
Description: Proportion of patients with both symptomatic remission and endoscopic healing at Week 10 (all individual IMU-838 doses were compared with one another and to placebo)
Time Frame: 10 weeks
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | 10 mg IMU-838 (Induction Phase) | 30 mg IMU-838 (Induction Phase) | 45 mg IMU-838 (Induction Phase) | Placebo (Induction Phase)
Number analyzed (Participants) | 62 | 56 | 60 | 57
Participants | 10 | 7 | 9 | 8

3. Secondary Outcome: Induction Phase: Symptomatic Remission
Description: Proportion of patients achieving symptomatic remission (Mayo rectal bleeding subscore = 0, and Mayo stool frequency subscore of 0 or 1) during the induction phase
Time Frame: 22 weeks
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Combined IMU-838 (30 or 45 mg IMU-838, Induction Phase) | Placebo (Induction Phase) | 10 mg IMU-838 (Induction Phase) | 30 mg IMU-838 (Induction Phase) | 45 mg IMU-838 (Induction Phase)
Number analyzed (Participants) | 128 | 62 | 66 | 64 | 64
Participants | 56 | 28 | 38 | 25 | 31

4. Secondary Outcome: Induction Phase: Time to Achieving Symptomatic Remission
Description: Time to achieving symptomatic remission (Mayo rectal bleeding subscore = 0 and Mayo stool frequency subscore of 0 or 1) within the extended induction phase
Time Frame: 22 weeks
Population: FAS
Measure: Mean (Standard Error); unit: days
Arm/Group | Combined IMU-838 (30 or 45 mg IMU-838, Induction Phase) | Placebo (Induction Phase) | 10 mg IMU-838 (Induction Phase) | 30 mg IMU-838 (Induction Phase) | 45 mg IMU-838 (Induction Phase)
Number analyzed (Participants) | 132 | 64 | 67 | 66 | 66
days | 108.8 (5.5) | 119.6 (7.1) | 98 (7.7) | 115.9 (7.4) | 101.9 (8.1)

5. Secondary Outcome: Induction Phase: Proportion of Patients With Clinical Response
Description: Proportion of patients with clinical response (decrease from Baseline in the full Mayo score of at least 3 points and at least 30%, with an accompanying decrease in the subscore for rectal bleeding of at least 1 point or an absolute subscore for rectal bleeding of 0 or 1) at Week 10
Time Frame: 10 weeks
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Combined IMU-838 (30 or 45 mg IMU-838, Induction Phase) | Placebo (Induction Phase) | 10 mg IMU-838 (Induction Phase) | 30 mg IMU-838 (Induction Phase) | 45 mg IMU-838 (Induction Phase)
Number analyzed (Participants) | 114 | 57 | 61 | 55 | 59
Participants | 50 | 27 | 31 | 23 | 27

6. Secondary Outcome: Induction Phase: Proportion of Patients With Endoscopic Healing
Description: Proportion of patients with endoscopic healing (Modified Mayo endoscopy subscore of 0 or 1) at Week 10
Time Frame: 10 weeks
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Combined IMU-838 (30 or 45 mg IMU-838, Induction Phase) | Placebo (Induction Phase) | 10 mg IMU-838 (Induction Phase) | 30 mg IMU-838 (Induction Phase) | 45 mg IMU-838 (Induction Phase)
Number analyzed (Participants) | 112 | 57 | 61 | 53 | 59
Participants | 28 | 12 | 18 | 14 | 14

7. Secondary Outcome: Induction Phase: Proportion of Patients With Symptomatic Response
Description: Proportion of patients with symptomatic response (≥1-point decrease from Baseline in Mayo PRO-2 score) during the induction phase (including extended induction phase)
Time Frame: 22 weeks
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Combined IMU-838 (30 or 45 mg IMU-838, Induction Phase) | Placebo (Induction Phase) | 10 mg IMU-838 (Induction Phase) | 30 mg IMU-838 (Induction Phase) | 45 mg IMU-838 (Induction Phase)
Number analyzed (Participants) | 128 | 62 | 66 | 64 | 64
Participants | 101 | 49 | 55 | 52 | 49

8. Secondary Outcome: Induction Phase: Full Mayo Score
Description: Change in full Mayo Score from Baseline to Week 10. The full Mayo score is composed of 4 categories (bleeding, stool frequency, physician assessment, and endoscopic appearance) each rated from 0 to 3 that are added up to give a total score that ranges from 0 to 12. A higher score indicates a worse outcome.
Time Frame: 10 weeks
Population: FAS
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Combined IMU-838 (30 or 45 mg IMU-838, Induction Phase) | Placebo (Induction Phase) | 10 mg IMU-838 (Induction Phase) | 30 mg IMU-838 (Induction Phase) | 45 mg IMU-838 (Induction Phase)
Number analyzed (Participants) | 132 | 64 | 67 | 66 | 66
score on a scale
  Baseline: number analyzed (Participants) | 131 | 64 | 67 | 65 | 66
  Baseline | 9.1 (1.4) | 9.1 (1.4) | 9.0 (1.6) | 9.1 (1.4) | 9.1 (1.4)
  Change from Baseline to Week 10: number analyzed (Participants) | 112 | 57 | 61 | 53 | 59
  Change from Baseline to Week 10 | -2.6 (2.7) | -2.3 (2.7) | -3.0 (2.6) | -2.5 (2.7) | -2.8 (2.7)

9. Secondary Outcome: Induction Phase: Partial Mayo Score
Description: Change in partial mayo score over 10 or 22 weeks. The partial Mayo score includes only the non-invasive Mayo subscores, ie, stool frequency, rectal bleeding, and physician's global assessment (each rated from 0 to 3 that are added up to give a total score that ranges from 0 to 9). A higher score indicates a worse outcome.
Time Frame: 22 weeks
Population: FAS
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Combined IMU-838 (30 or 45 mg IMU-838, Induction Phase) | Placebo (Induction Phase) | 10 mg IMU-838 (Induction Phase) | 30 mg IMU-838 (Induction Phase) | 45 mg IMU-838 (Induction Phase)
Number analyzed (Participants) | 132 | 64 | 67 | 66 | 66
score on a scale
  Baseline (all patients): number analyzed (Participants) | 131 | 64 | 67 | 65 | 66
  Baseline (all patients) | 6.6 (1.2) | 6.5 (1.1) | 6.4 (1.4) | 6.5 (1.2) | 6.6 (1.2)
  Change from Baseline to Week 10 (all patients): number analyzed (Participants) | 117 | 58 | 62 | 56 | 61
  Change from Baseline to Week 10 (all patients) | -2.2 (2.2) | -1.9 (2.2) | -2.4 (2.2) | -1.9 (2.0) | -2.4 (2.3)
  Baseline (only patients who entered extended induction phase): number analyzed (Participants) | 47 | 27 | 28 | 24 | 23
  Baseline (only patients who entered extended induction phase) | 6.6 (1.2) | 6.5 (1.0) | 6.6 (1.3) | 6.6 (1.2) | 6.7 (1.2)
  Change from Baseline to Week 22 (only patients who entered extended induction phase): number analyzed (Participants) | 45 | 27 | 27 | 23 | 22
  Change from Baseline to Week 22 (only patients who entered extended induction phase) | -3.5 (2.1) | -3.6 (2.2) | -3.4 (2.3) | -3.7 (2.2) | -3.3 (2.0)

10. Secondary Outcome: Induction Phase: Patient Reported Outcome (PRO)-2 Mayo Score
Description: Change in PRO-2 Mayo score over 10 or 22 weeks. Mayo PRO-2 score, ie, stool frequency and rectal bleeding score each rated from 0 to 3 that are added up to give a total score that ranges from 0 to 6. A higher score indicates a worse outcome.
Time Frame: 22 weeks
Population: FAS
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Combined IMU-838 (30 or 45 mg IMU-838, Induction Phase) | Placebo (Induction Phase) | 10 mg IMU-838 (Induction Phase) | 30 mg IMU-838 (Induction Phase) | 45 mg IMU-838 (Induction Phase)
Number analyzed (Participants) | 132 | 64 | 67 | 66 | 66
score on a scale
  Baseline (all patients): number analyzed (Participants) | 131 | 64 | 67 | 65 | 66
  Baseline (all patients) | 4.3 (1.0) | 4.3 (0.9) | 4.1 (1.2) | 4.3 (1.0) | 4.3 (1.0)
  Change from Baseline to Week 10 (all patients): number analyzed (Participants) | 117 | 58 | 62 | 56 | 61
  Change from Baseline to Week 10 (all patients) | -1.6 (1.7) | -1.4 (1.7) | -1.7 (1.6) | -1.4 (1.6) | -1.8 (1.7)
  Baseline (only patients who entered extended induction phase): number analyzed (Participants) | 47 | 27 | 28 | 24 | 23
  Baseline (only patients who entered extended induction phase) | 4.3 (1.0) | 4.3 (0.8) | 4.2 (1.1) | 4.3 (1.1) | 4.3 (1.0)
  Change from Baseline to Week 22 (only patients who entered extended induction phase): number analyzed (Participants) | 43 | 27 | 27 | 21 | 22
  Change from Baseline to Week 22 (only patients who entered extended induction phase) | -2.5 (1.6) | -2.6 (1.6) | -2.4 (1.8) | -2.7 (1.6) | -2.3 (1.6)

11. Secondary Outcome: Induction Phase: Fecal Calprotectin (fCP)
Description: Time course of biomarker fCP in stool samples during extended induction phase
Time Frame: 22 weeks
Population: FAS
Measure: Median (Full Range); unit: mg/kg
Arm/Group | Combined IMU-838 (30 or 45 mg IMU-838, Induction Phase) | Placebo (Induction Phase) | 10 mg IMU-838 (Induction Phase) | 30 mg IMU-838 (Induction Phase) | 45 mg IMU-838 (Induction Phase)
Number analyzed (Participants) | 132 | 64 | 67 | 66 | 66
mg/kg
  Day 0 (all patients): number analyzed (Participants) | 113 | 54 | 58 | 56 | 57
  Day 0 (all patients) | 799.0 [9 to 10437] | 899.0 [39 to 5323] | 697.0 [3 to 4064] | 711.5 [55 to 10437] | 992.0 [9 to 8310]
  Week 10 (all patients: number analyzed (Participants) | 90 | 50 | 48 | 44 | 46
  Week 10 (all patients | 290.0 [13 to 6731] | 405.0 [9 to 17819] | 384.0 [3 to 19955] | 301.5 [13 to 5269] | 265.0 [17 to 6731]
  Day 0 (Only patients who entered extended induction phase): number analyzed (Participants) | 38 | 20 | 25 | 18 | 20
  Day 0 (Only patients who entered extended induction phase) | 616.5 [9 to 10437] | 1039.0 [46 to 5323] | 603.0 [60 to 2536] | 547.0 [115 to 10437] | 856.5 [9 to 8310]
  Week 22 (Only patients who entered extended induction phase): number analyzed (Participants) | 29 | 26 | 16 | 14 | 15
  Week 22 (Only patients who entered extended induction phase) | 332.0 [6 to 6699] | 387.0 [38 to 4183] | 353.0 [20 to 1515] | 314.0 [6 to 1124] | 576.0 [16 to 6699]

12. Secondary Outcome: Induction Phase: C-reactive Protein (CRP)
Description: Time course of biomarker CRP in blood samples during extended induction phase
Time Frame: 22 weeks
Population: FAS
Measure: Median (Full Range); unit: mg/L
Arm/Group | Combined IMU-838 (30 or 45 mg IMU-838, Induction Phase) | Placebo (Induction Phase) | 10 mg IMU-838 (Induction Phase) | 30 mg IMU-838 (Induction Phase) | 45 mg IMU-838 (Induction Phase)
Number analyzed (Participants) | 132 | 64 | 67 | 66 | 66
mg/L
  Day 0 (all patients): number analyzed (Participants) | 131 | 64 | 67 | 66 | 65
  Day 0 (all patients) | 3.50 [0.3 to 122.3] | 3.2 [0.3 to 81.1] | 5.30 [0.3 to 79.8] | 3.70 [0.3 to 122.3] | 3.50 [0.3 to 80.0]
  Week 10 (all patients): number analyzed (Participants) | 106 | 56 | 59 | 52 | 54
  Week 10 (all patients) | 3.40 [0.3 to 33.9] | 1.85 [0.3 to 50.8] | 4.00 [0.3 to 46.0] | 3.50 [0.3 to 26.3] | 2.75 [0.3 to 33.9]
  Day 0 (Only patients who entered extended induction phase): number analyzed (Participants) | 46 | 27 | 28 | 24 | 22
  Day 0 (Only patients who entered extended induction phase) | 3.65 [0.3 to 113.8] | 2.40 [0.3 to 78.6] | 5.55 [0.3 to 61.4] | 3.05 [0.3 to 113.8] | 7.85 [0.3 to 80.0]
  Week 22 (Only patients who entered extended induction phase): number analyzed (Participants) | 33 | 26 | 21 | 17 | 16
  Week 22 (Only patients who entered extended induction phase) | 2.70 [0.3 to 23.7] | 1.25 [0.3 to 69.9] | 2.80 [0.3 to 17.8] | 2.00 [0.3 to 13.0] | 2.75 [0.3 to 23.7]

13. Secondary Outcome: Safety: Adverse Events
Description: Incidence and Severity of AEs during the induction and maintenance phases
Time Frame: 50 weeks
Population: SAF
Measure: Count of Participants; unit: Participants
Groups:
- 10 mg IMU-838 (Maintenance Phase: Two 5 mg tablets once daily of IMU-838 for up to 40 weeks.
- 30 mg IMU-838 (Maintenance Phase): Two 15 mg tablets once daily of IMU-838 for up to 40 weeks.
Arm/Group | 10 mg IMU-838 (Induction Phase) | 30 mg IMU-838 (Induction Phase) | 45 mg IMU-838 (Induction Phase) | Placebo (Induction Phase) | 10 mg IMU-838 (Maintenance Phase | 30 mg IMU-838 (Maintenance Phase) | Placebo (Maintenance Phase)
Number analyzed (Participants) | 67 | 67 | 66 | 63 | 45 | 40 | 27
Participants
  Any TEAE | 28 | 30 | 30 | 23 | 16 | 16 | 12
  Any mild TEAE | 23 | 21 | 24 | 15 | 11 | 12 | 8
  Any moderate TEAE | 7 | 10 | 11 | 13 | 5 | 7 | 4
  Any severe TEAE | 2 | 3 | 2 | 0 | 2 | 2 | 0

14. Secondary Outcome: Safety: Number of Participants With Clinically Significant Findings During Physical Examination
Description: The emergence of any clinically significant findings compared to screening captured during the induction and maintenance phases
Time Frame: 50 weeks
Population: SAF
Measure: Count of Participants; unit: Participants
Groups:
- 10 mg IMU-838 (Maintenace Phase): Two 5 mg tablets once daily of IMU-838 for up to 40 weeks.
Arm/Group | 10 mg IMU-838 (Induction Phase) | 30 mg IMU-838 (Induction Phase) | 45 mg IMU-838 (Induction Phase) | Placebo (Induction Phase) | 10 mg IMU-838 (Maintenace Phase) | 30 mg IMU-383 (Maintenance Phase) | Placebo (Maintenance Phase)
Number analyzed (Participants) | 67 | 67 | 66 | 63 | 45 | 40 | 27
Participants | 0 | 3 | 4 | 0 | 2 | 1 | 2

15. Secondary Outcome: Safety: Body Weight
Description: Changes in body weight during the induction and maintenance phases
Time Frame: 50 weeks
Population: SAF
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | 10 mg IMU-838 (Induction Phase) | 30 mg IMU-838 (Induction Phase) | 45 mg IMU-838 (Induction Phase) | Placebo (Induction Phase) | 10 mg IMU-838 (Maintenance Phase | 30 mg IMU-838 (Maintenance Phase) | Placebo (Maintenance Phase)
Number analyzed (Participants) | 67 | 67 | 66 | 63 | 45 | 40 | 27
kg
  Induction phase - Day 0: number analyzed (Participants) | 67 | 67 | 66 | 63 | 0 | 0 | 0
  Induction phase - Day 0 | 73.881 (19.479) | 72.436 (15.348) | 73.959 (13.915) | 70.141 (15.754) |  |  |
  Induction phase - Week 10: number analyzed (Participants) | 58 | 54 | 54 | 55 | 0 | 0 | 0
  Induction phase - Week 10 | 73.747 (20.030) | 71.457 (14.522) | 75.094 (14.148) | 71.437 (15.998) |  |  |
  Induction phase - Week 22: number analyzed (Participants) | 22 | 18 | 17 | 26 | 0 | 0 | 0
  Induction phase - Week 22 | 70.310 (13.640) | 74.689 (15.143) | 75.188 (18.202) | 69.635 (14.425) |  |  |
  Maintenance phase - Baseline: number analyzed (Participants) | 0 | 0 | 0 | 0 | 45 | 40 | 27
  Maintenance phase - Baseline |  |  |  |  | 74.431 (13.081) | 70.490 (16.480) | 72.441 (13.259)
  Maintenance phase - Week 50: number analyzed (Participants) | 0 | 0 | 0 | 0 | 34 | 29 | 21
  Maintenance phase - Week 50 |  |  |  |  | 75.743 (13.452) | 73.986 (18.069) | 70.310 (11.458)

16. Secondary Outcome: Safety: Blood Pressure
Description: Changes in blood pressure (mm Hg) during the induction and maintenance phases
Time Frame: 50 weeks
Population: SAF
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | 10 mg IMU-838 (Induction Phase) | 30 mg IMU-838 (Induction Phase) | 45 mg IMU-838 (Induction Phase) | Placebo (Induction Phase) | 10 mg IMU-838 (Maintenance Phase) | 30 mg IMU-838 (Maintenance Phase) | Placebo (Maintenance Phase)
Number analyzed (Participants) | 67 | 67 | 66 | 63 | 45 | 40 | 27
mmHg
  Induction phase - Day 0 (systolic blood pressure): number analyzed (Participants) | 67 | 67 | 66 | 63 | 0 | 0 | 0
  Induction phase - Day 0 (systolic blood pressure) | 123.2 (14.2) | 125.1 (12.8) | 123.2 (11.4) | 121.9 (11.8) |  |  |
  Induction phase - Week 10 (systolic blood pressure): number analyzed (Participants) | 59 | 54 | 54 | 55 | 0 | 0 | 0
  Induction phase - Week 10 (systolic blood pressure) | 123.1 (11.4) | 123.8 (13.2) | 121.7 (9.7) | 122.0 (12.8) |  |  |
  Induction phase - Week 22 (systolic blood pressure): number analyzed (Participants) | 22 | 18 | 17 | 26 | 0 | 0 | 0
  Induction phase - Week 22 (systolic blood pressure) | 118.3 (10.2) | 126.7 (12.3) | 119.8 (6.6) | 121.8 (12.3) |  |  |
  Induction phase - Day 0 (diastolic blood pressure): number analyzed (Participants) | 67 | 67 | 66 | 63 | 0 | 0 | 0
  Induction phase - Day 0 (diastolic blood pressure) | 76.2 (10.8) | 78.1 (10.3) | 79.5 (9.4) | 74.9 (8.2) |  |  |
  Induction phase - Week 10 (diastolic blood pressure): number analyzed (Participants) | 59 | 54 | 54 | 55 | 0 | 0 | 0
  Induction phase - Week 10 (diastolic blood pressure) | 76.1 (9.1) | 79.5 (9.2) | 77.3 (7.9) | 75.5 (7.9) |  |  |
  Induction phase - Week 22 (diastolic blood pressure): number analyzed (Participants) | 22 | 18 | 17 | 26 | 0 | 0 | 0
  Induction phase - Week 22 (diastolic blood pressure) | 72.0 (7.6) | 77.6 (7.4) | 75.4 (6.5) | 74.2 (9.8) |  |  |
  Maintenance phase - baseline (systolic blood pressure): number analyzed (Participants) | 0 | 0 | 0 | 0 | 45 | 40 | 27
  Maintenance phase - baseline (systolic blood pressure) |  |  |  |  | 121.3 (10.6) | 123.7 (12.2) | 124.1 (13.0)
  Maintenance phase - Week 50 (systolic blood pressure): number analyzed (Participants) | 0 | 0 | 0 | 0 | 34 | 29 | 21
  Maintenance phase - Week 50 (systolic blood pressure) |  |  |  |  | 122.0 (13.0) | 125.3 (14.3) | 122.6 (9.2)
  Maintenance phase - baseline (diastolic blood pressure): number analyzed (Participants) | 0 | 0 | 0 | 0 | 45 | 40 | 27
  Maintenance phase - baseline (diastolic blood pressure) |  |  |  |  | 75.2 (8.7) | 76.5 (9.5) | 75.1 (8.8)
  Maintenance phase - Week 50 (diastolic blood pressure: number analyzed (Participants) | 0 | 0 | 0 | 0 | 34 | 29 | 21
  Maintenance phase - Week 50 (diastolic blood pressure |  |  |  |  | 76.5 (9.9) | 77.1 (9.0) | 74.7 (6.4)

17. Secondary Outcome: Safety: Heart Rate
Description: Changes in heart rate (beats per minute) during the induction and maintenance phases
Time Frame: 50 weeks
Population: SAF
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | 10 mg IMU-838 (Induction Phase) | 30 mg IMU-838 (Induction Phase) | 45 mg IMU-838 (Induction Phase) | Placebo (Induction Phase) | 10 mg IMU-838 (Maintenance Phase) | 30 mg IMU-838 (Maintenance Phase) | Placebo (Maintenance Phase)
Number analyzed (Participants) | 67 | 67 | 66 | 63 | 45 | 40 | 27
beats per minute
  Induction phase - Day 0: number analyzed (Participants) | 67 | 67 | 66 | 63 | 0 | 0 | 0
  Induction phase - Day 0 | 74.7 (13.6) | 77.4 (12.3) | 73.6 (8.9) | 73.5 (9.0) |  |  |
  Induction phase - Week 10: number analyzed (Participants) | 59 | 54 | 54 | 55 | 0 | 0 | 0
  Induction phase - Week 10 | 76.1 (13.9) | 74.1 (10.4) | 73.6 (9.0) | 73.9 (10.8) |  |  |
  Induction phase - Week 22: number analyzed (Participants) | 22 | 18 | 17 | 26 | 0 | 0 | 0
  Induction phase - Week 22 | 69.6 (13.0) | 71.9 (9.1) | 71.6 (6.2) | 70.8 (7.1) |  |  |
  Maintenance phase -Baseline: number analyzed (Participants) | 0 | 0 | 0 | 0 | 45 | 40 | 27
  Maintenance phase -Baseline |  |  |  |  | 73.0 (9.2) | 73.4 (7.5) | 72.4 (9.7)
  Maintenance phase - Week 50: number analyzed (Participants) | 0 | 0 | 0 | 0 | 34 | 29 | 21
  Maintenance phase - Week 50 |  |  |  |  | 73.0 (8.6) | 73.2 (6.5) | 75.4 (10.7)

18. Secondary Outcome: Safety: 12-lead Electrocardiogram (ECG)
Description: Number of patients with clinically significant changes in ECG
Time Frame: 50 weeks
Population: SAF
Measure: Count of Participants; unit: Participants
Arm/Group | 10 mg IMU-838 (Induction Phase) | 30 mg IMU-838 (Induction Phase) | 45 mg IMU-838 (Induction Phase) | Placebo (Induction Phase) | 10 mg IMU-838 (Maintenance Phase) | 30 mg IMU-838 (Maintenance Phase) | Placebo (Maintenance Phase)
Number analyzed (Participants) | 67 | 67 | 66 | 63 | 45 | 40 | 27
Participants | 0 | 1 | 0 | 0 | 0 | 0 | 0

19. Secondary Outcome: Safety: Hematology
Description: Number of participants with abnormal hematology laboratory values (treatment-emergent adverse events [TEAEs] related to hematological abnormalities)
Time Frame: up to Week 50
Population: SAF
Measure: Count of Participants; unit: Participants
Arm/Group | 10 mg IMU-838 (Induction Phase) | 30 mg IMU-838 (Induction Phase) | 45 mg IMU-838 (Induction Phase) | Placebo (Induction Phase) | 10 mg IMU-838 (Maintenance Phase | 30 mg IMU-838 (Maintenance Phase) | Placebo (Maintenance Phase)
Number analyzed (Participants) | 67 | 67 | 66 | 63 | 45 | 40 | 27
Participants
  Anemia | 3 | 6 | 4 | 3 | 1 | 2 | 2
  Leukopenia | 1 | 1 | 0 | 0 | 0 | 0 | 0
  Neutropenia | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Thrombocytosis | 0 | 1 | 0 | 1 | 0 | 0 | 1
  Hemoglobin decreased | 0 | 2 | 9 | 0 | 1 | 0 | 0
  Platelet count increased | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Leukocytosis | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Microcytic anemia | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Neutrophil count increased | 0 | 0 | 0 | 0 | 0 | 0 | 1
  White blood cell count increased | 0 | 0 | 0 | 0 | 0 | 0 | 1

20. Secondary Outcome: Safety: Blood Chemistry
Description: Number of participants with abnormal blood chemistry laboratory values (TEAES related to clinical chemistry abnormalities)
Time Frame: 50 weeks
Population: SAF
Measure: Count of Participants; unit: Participants
Arm/Group | 10 mg IMU-838 (Induction Phase) | 30 mg IMU-838 (Induction Phase) | 45 mg IMU-838 (Induction Phase) | Placebo (Induction Phase) | 10 mg IMU-838 (Maintenance Phase) | 30 mg IMU-383 (Maintenance Phase) | Placebo (Maintenance Phase)
Number analyzed (Participants) | 67 | 67 | 66 | 63 | 45 | 40 | 27
Participants
  Alanine transferase increased | 2 | 0 | 0 | 1 | 0 | 0 | 0
  Amylase increased | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Aspartate aminotransferase increased | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Blood bilirubin increased | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Blood bilirubin unconjugated increased | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Blood calcium decreased | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Blood cholesterol increased | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Blood creatinine increased | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Blood creatine phosphokinase MB increased | 1 | 1 | 0 | 0 | 0 | 0 | 0
  Blood creatine phosphokinase increased | 1 | 2 | 0 | 0 | 0 | 0 | 1
  Blood potassium increased | 1 | 0 | 1 | 1 | 0 | 0 | 0
  Blood triglycerides increased | 0 | 1 | 0 | 1 | 0 | 0 | 0
  C-reactive protein increased | 0 | 2 | 1 | 0 | 0 | 0 | 0
  Fecal calprotectin increased | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Gamma-glutamyltransferase increased | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Hepatic enzyme increased | 0 | 0 | 1 | 1 | 0 | 0 | 1
  Hyperbilirubinemia | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Hyperkalemia | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Hyperlipasemia | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Hypertriglyceridemia | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Hyperuricemia | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Hypokalemia | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Hypophosphatasemia | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Liver function test abnormal | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Lipase increased | 0 | 0 | 0 | 0 | 1 | 1 | 1

21. Secondary Outcome: Safety: Coagulation
Description: Number of participants with clinically significant abnormal coagulation laboratory values
Time Frame: 10 weeks
Population: SAF, Coagulation parameters were only analyzed in the Induction phase.
Measure: Count of Participants; unit: Participants
Arm/Group | 10 mg IMU-838 (Induction Phase) | 30 mg IMU-838 (Induction Phase) | 45 mg IMU-838 (Induction Phase) | Placebo (Induction Phase)
Number analyzed (Participants) | 67 | 67 | 66 | 63
Participants | 0 | 0 | 0 | 0

22. Secondary Outcome: Safety: Urinalysis
Description: Number of participants with abnormal urinalysis laboratory values (TEAEs related to urinalysis)
Time Frame: 50 weeks
Population: SAF
Measure: Count of Participants; unit: Participants
Arm/Group | 10 mg IMU-838 (Induction Phase) | 30 mg IMU-838 (Induction Phase) | 45 mg IMU-838 (Induction Phase) | Placebo (Induction Phase) | 10 mg IMU-838 (Maintenance Phase) | 30 mg IMU-838 (Maintenance Phase) | Placebo (Maintenance Phase)
Number analyzed (Participants) | 67 | 67 | 66 | 63 | 45 | 40 | 27
Participants
  Blood urine present | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Creatinine urine increased | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Crystalluria | 0 | 2 | 0 | 0 | 0 | 0 | 0
  Hematuria | 0 | 0 | 5 | 1 | 0 | 2 | 0
  Hemorrhage urinary tract | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Hyperoxaluria | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Hyperuricosuria | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Ketonuria | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Micturition urgency | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Proteinuria | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Red blood cells urine positive | 0 | 1 | 1 | 0 | 0 | 0 | 1
  Renal colic | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Renal Cyst | 0 | 1 | 0 | 0 | 0 | 0 | 0

23. Secondary Outcome: Safety: Micro Ribonucleic Acid-122 Expression
Description: Micro ribonucleic acid-122 (miR-122) expression (before first dose and 24 hours after first dose - foldchange of normalized expression values )
Time Frame: 24 hours
Population: SAF
Measure: Mean (Standard Deviation); unit: fold change
Arm/Group | 10 mg IMU-838 (Induction Phase) | 30 mg IMU-838 (Induction Phase) | 45 mg IMU-838 (Induction Phase) | Placebo (Induction Phase)
Number analyzed (Participants) | 61 | 60 | 59 | 60
fold change | 2.0276 (2.7747) | 3.5573 (10.8852) | 1.8842 (3.5346) | 2.5739 (5.2723)

24. Secondary Outcome: Pharmacodynamics (PK): IMU-838 Trough Level
Description: Measurement of pre-dose (trough) blood plasma levels of IMU-838 throughout the induction period
Time Frame: Day 0, Day 1, Day 7, Week 2 and Week 10
Population: SAF
Measure: Median (Full Range); unit: µg/mL
Arm/Group | 10 mg IMU-838 (Induction Phase) | 30 mg IMU-838 (Induction Phase) | 45 mg IMU-838 (Induction Phase)
Number analyzed (Participants) | 67 | 67 | 66
µg/mL
  Day 0: number analyzed (Participants) | 57 | 62 | 59
  Day 0 | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 7.34] | 0.00 [0.00 to 0.00]
  Day 1: number analyzed (Participants) | 56 | 62 | 59
  Day 1 | 0.30 [0.00 to 1.74] | 0.94 [0.00 to 3.75] | 1.41 [0.00 to 5.63]
  Day 7: number analyzed (Participants) | 63 | 62 | 60
  Day 7 | 0.58 [0.00 to 2.13] | 1.71 [0.00 to 8.82] | 2.77 [0.70 to 8.29]
  Week 2: number analyzed (Participants) | 58 | 58 | 59
  Week 2 | 0.97 [0.00 to 3.00] | 3.24 [0.00 to 8.54] | 5.23 [1.30 to 11.0]
  Week 10: number analyzed (Participants) | 53 | 48 | 50
  Week 10 | 1.17 [0.00 to 3.43] | 3.32 [0.00 to 9.32] | 5.03 [0.93 to 11.80]

25. Secondary Outcome: PK: IMU-838 Plasma Level
Description: Measurement of post-dose blood plasma levels of IMU-838 at Week 2
Time Frame: 2 weeks
Population: SAF
Measure: Median (Full Range); unit: µg/mL
Arm/Group | 10 mg IMU-838 (Induction Phase) | 30 mg IMU-838 (Induction Phase) | 45 mg IMU-838 (Induction Phase)
Number analyzed (Participants) | 58 | 63 | 58
µg/mL | 2.30 [0.00 to 4.23] | 6.05 [0.00 to 12.40] | 10.70 [1.68 to 23.40]

26. Secondary Outcome: PK: Area Under the Drug Concentration-time Curve (AUC) From Time Zero to 24 Hours (AUC0-24h)
Description: Single-dose PK measurement of AUC0-24h in a subset of patients in the open-label phase
Time Frame: pre-dose, 1, 2, 3, 4, 5, 6 hours post PK dose; 24 hours post PK dose; 48 hours post PK dose; 72 hours post PK dose
Population: No data were collected for this endpoint.
Arm/Group | 30 mg IMU-838 (Open-label Phase)
Number analyzed (Participants) | 0

27. Secondary Outcome: PK: AUC Time Zero to Last Measurable Concentration (AUC0-t)
Description: Single-dose PK measurement of AUC0-t in a subset of patients in the open-label phase
Time Frame: pre-dose, 1, 2, 3, 4, 5, 6 hours post PK dose; 24 hours post PK dose; 48 hours post PK dose; 72 hours post PK dose
Population: No data were collected for this endpoint.
Arm/Group | 30 mg IMU-838 (Open-label Phase)
Number analyzed (Participants) | 0

28. Secondary Outcome: PK: AUC Time Zero to Infinity (AUC0-inf)
Description: Single-dose PK measurement of AUC0-inf in a subset of patients in the open-label phase
Time Frame: pre-dose, 1, 2, 3, 4, 5, 6 hours post PK dose; 24 hours post PK dose; 48 hours post PK dose; 72 hours post PK dose
Population: No data were collected for this endpoint.
Arm/Group | 30 mg IMU-838 (Open-label Phase)
Number analyzed (Participants) | 0

29. Secondary Outcome: PK: Maximum Plasma Concentration (Cmax)
Description: Single-dose PK measurement of Cmax in a subset of patients in the open-label phase
Time Frame: pre-dose, 1, 2, 3, 4, 5, 6 hours post PK dose; 24 hours post PK dose; 48 hours post PK dose; 72 hours post PK dose
Population: No data were collected for this endpoint.
Arm/Group | 30 mg IMU-838 (Open-label Phase)
Number analyzed (Participants) | 0

30. Secondary Outcome: PK: Time to Cmax (Tmax)
Description: Single-dose PK measurement of Tmax in a subset of patients in the open-label phase
Time Frame: pre-dose, 1, 2, 3, 4, 5, 6 hours post PK dose; 24 hours post PK dose; 48 hours post PK dose; 72 hours post PK dose
Population: No data were collected for this endpoint.
Arm/Group | 30 mg IMU-838 (Open-label Phase)
Number analyzed (Participants) | 0

31. Secondary Outcome: Maintenance Phase: Proportion of Patients in Symptomatic Remission
Description: Proportion of patients in symptomatic remission (Mayo rectal bleeding subscore = 0, and Mayo stool frequency subscore of 0 or 1) by visit up to Week 50 in maintenance phase
Time Frame: Week 14, Week 30, Week 50
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | 10 mg IMU-838 (Maintenance Phase) | 30 mg IMU-838 (Maintenance Phase) | Placebo (Maintenance Phase)
Number analyzed (Participants) | 45 | 40 | 27
Participants
  Week 14: number analyzed (Participants) | 19 | 20 | 11
  Week 14 | 16 | 14 | 7
  Week 30: number analyzed (Participants) | 40 | 33 | 24
  Week 30 | 33 | 23 | 19
  Week 50: number analyzed (Participants) | 33 | 29 | 21
  Week 50 | 27 | 24 | 16

32. Secondary Outcome: Maintenance Phase: Mayo PRO-2 Score
Description: Time course of Mayo PRO-2 score until Week 50. Mayo patient-reported outcome score, ie, stool frequency and rectal bleeding score each rated from 0 to 3 3 that are added up to give a total score that ranges from 0 to 6. A higher score indicates a worse outcome.
Time Frame: 50 weeks
Population: FAS
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 10 mg IMU-838 (Maintenance Phase) | 30 mg IMU-838 (Maintenance Phase) | Placebo (Maintenance Phase)
Number analyzed (Participants) | 45 | 40 | 27
score on a scale
  Maintenance phase Baseline | 0.8 (0.5) | 0.9 (0.8) | 0.7 (0.5)
  Change from Baseline to Week 50: number analyzed (Participants) | 33 | 29 | 21
  Change from Baseline to Week 50 | 0.1 (0.9) | 0.2 (1.1) | 0.4 (0.9)

33. Secondary Outcome: Maintenance Phase: Time to Relapse
Description: Time to symptomatic ulcerative colitis (UC) relapse
Time Frame: 50 weeks
Population: FAS
Measure: Mean (Standard Error); unit: days
Arm/Group | 10 mg IMU-838 (Maintenance Phase) | 30 mg IMU-838 (Maintenance Phase) | Placebo (Maintenance Phase)
Number analyzed (Participants) | 45 | 40 | 27
days | 231.7 (10) | 221.9 (16.2) | 186.6 (10.2)

34. Secondary Outcome: Maintenance Phase: Proportion of Patients Without Relapse
Description: Proportion of patients without symptomatic UC relapse until Week 50
Time Frame: 50 weeks
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | 10 mg IMU-838 (Maintenance Phase) | 30 mg IMU-838 (Maintenance Phase) | Placebo (Maintenance Phase)
Number analyzed (Participants) | 43 | 36 | 26
Participants | 32 | 24 | 18

35. Secondary Outcome: Maintenance Phase: fCP
Description: Timecourse of biomarker fCP in stool samples
Time Frame: 50 weeks
Population: FAS
Measure: Median (Full Range); unit: mg/kg
Arm/Group | 10 mg IMU-838 (Maintenance Phase) | 30 mg IMU-838 (Maintenance Phase) | Placebo (Maintenance Phase)
Number analyzed (Participants) | 45 | 40 | 27
mg/kg
  Maintenance phase Baseline: number analyzed (Participants) | 44 | 40 | 27
  Maintenance phase Baseline | 256.5 [3 to 1948] | 207.0 [3 to 16359] | 335.0 [9 to 4183]
  Week 14: number analyzed (Participants) | 17 | 19 | 11
  Week 14 | 99.0 [16 to 611] | 145.0 [12 to 2386] | 353.0 [19 to 2529]
  Week 30: number analyzed (Participants) | 33 | 31 | 21
  Week 30 | 149.0 [3 to 3169] | 217.0 [22 to 2431] | 210.0 [2 to 1694]
  Week 50: number analyzed (Participants) | 27 | 19 | 17
  Week 50 | 181.0 [11 to 1931] | 147.0 [27 to 5777] | 364.0 [18 to 1617]

36. Secondary Outcome: Maintenance Phase: CRP
Description: Timecourse of biomarker CRP in blood samples
Time Frame: 50 weeks
Population: FAS
Measure: Median (Full Range); unit: mg/L
Arm/Group | 10 mg IMU-838 (Maintenance Phase) | 30 mg IMU-838 (Maintenance Phase) | Placebo (Maintenance Phase)
Number analyzed (Participants) | 45 | 40 | 27
mg/L
  Maintenance phase Baseline | 1.30 [0.3 to 105.7] | 2.50 [0.3 to 38.2] | 1.10 [0.3 to 5.2]
  Week 14: number analyzed (Participants) | 19 | 21 | 11
  Week 14 | 1.10 [0.3 to 19.2] | 1.50 [0.3 to 23.4] | 1.90 [0.3 to 7.6]
  Week 30: number analyzed (Participants) | 36 | 34 | 22
  Week 30 | 1.30 [0.3 to 48.3] | 2.05 [0.3 to 172.3] | 1.00 [0.3 to 21.0]
  Week 50: number analyzed (Participants) | 27 | 24 | 18
  Week 50 | 1.10 [0.3 to 12.2] | 3.60 [0.3 to 56.0] | 1.95 [0.3 to 18.6]

37. Secondary Outcome: Maintenance Phase: Proportion of Patients With Endoscopic Healing
Description: Proportion of patients with endoscopic healing (Modified Mayo endoscopy subscore of 0 or 1) at Week 50 of maintenance phase
Time Frame: 50 weeks
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | 10 mg IMU-838 (Maintenance Phase) | 30 mg IMU-838 (Maintenance Phase) | Placebo (Maintenance Phase)
Number analyzed (Participants) | 28 | 26 | 17
Participants | 15 | 19 | 6

38. Secondary Outcome: Maintenance Phase: Proportion of Patients With Microscopic Healing
Description: Proportion of patients with microscopic healing (Geboes score of =< 3.1) at Week 50 of maintenance phase
Time Frame: 50 weeks
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | 10 mg IMU-838 (Maintenance Phase) | 30 mg IMU-838 (Maintenance Phase) | Placebo (Maintenance Phase)
Number analyzed (Participants) | 30 | 26 | 17
Participants | 25 | 20 | 12

39. Secondary Outcome: Maintenance Phase: Corticosteroid-free Remission
Description: Corticosteroid-free clinical remission (clinical remission and no receipt of systemic or local corticosteroids) at Week 50 in patients receiving corticosteroids at Baseline
Time Frame: 50 weeks
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | 10 mg IMU-838 (Maintenance Phase) | 30 mg IMU-838 (Maintenance Phase) | Placebo (Maintenance Phase)
Number analyzed (Participants) | 26 | 26 | 18
Participants | 10 | 16 | 5

40. Secondary Outcome: Open-label Phase: Symptom Control
Description: Proportion of patients with symptom control
Time Frame: up to 4 years
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | 30 mg IMU-838 (Open-label Phase)
Number analyzed (Participants) | 190
Participants | 55

41. Secondary Outcome: Open-label Phase: fCP
Description: Timecourse of biomarker fCP in stool samples. Visits were scheduled every 4 weeks (+/-7 days) until 50 weeks of total study participation (ie induction + extended induction, if applicable, maintenance + open-label part) and every 10 weeks (+/-7 days) thereafter. The visit schedule in the OLE after 50 weeks of overall study treatment was changed from a 10-week schedule to a 24 week (+/-14 days) schedule after Protocol Version 6.0 came into force.
  Because the study was terminated early, EoT varied between patients depending on when patients entered the study and the time a patient participated in the induction and maintenance phases before switching to the OLE.
Time Frame: Baseline, Week 4 OLE, Week 8 OLE, EoT up to 4 years (variable)
Population: FAS, separated by entry in OLE, data only shown if number of patients included in analysis ≥ 5 per visit
Measure: Median (Full Range); unit: mg/kg
Arm/Group | 30 mg IMU-838 (Open-label Phase)
Number analyzed (Participants) | 190
mg/kg
  Entry in OLE after (extended) induction phase - Baseline: number analyzed (Participants) | 111
  Entry in OLE after (extended) induction phase - Baseline | 542.0 [6 to 19955]
  Entry in OLE after (extended) induction phase - Visit 1 (Week 4 OLE): number analyzed (Participants) | 8
  Entry in OLE after (extended) induction phase - Visit 1 (Week 4 OLE) | 557.0 [98 to 4774]
  Entry in OLE after (extended) induction phase - Visit 2 (Week 8 OLE): number analyzed (Participants) | 7
  Entry in OLE after (extended) induction phase - Visit 2 (Week 8 OLE) | 467.0 [55 to 2271]
  Entry in OLE after (extended) induction phase - end of treatment (up to 4 years, variable): number analyzed (Participants) | 53
  Entry in OLE after (extended) induction phase - end of treatment (up to 4 years, variable) | 234.0 [5 to 9906]
  Entry in OLE after maintenance phase - Baseline: number analyzed (Participants) | 75
  Entry in OLE after maintenance phase - Baseline | 221.0 [8 to 5777]
  Entry in OLE after maintenance phase - end of treatment (up to 4 years, variable): number analyzed (Participants) | 43
  Entry in OLE after maintenance phase - end of treatment (up to 4 years, variable) | 168.0 [3 to 5256]

42. Secondary Outcome: Open-label Phase: CRP
Description: Timecourse of biomarker CRP in blood samples. Visits were scheduled every 4 weeks (+/-7 days) until 50 weeks of total study participation (ie induction + extended induction, if applicable, maintenance + open-label part) and every 10 weeks (+/-7 days) thereafter. The visit schedule in the OLE after 50 weeks of overall study treatment was changed from a 10-week schedule to a 24 week (+/-14 days) schedule after Protocol Version 6.0 came into force.
  Because the study was terminated early, EoT varied between patients depending on when patients entered the study and the time a patient participated in the induction and maintenance phases before switching to the OLE.
Time Frame: Baseline, Week 4 OLE, Week 8 OLE, Week 10 OLE, Week 12 OLE, Week 16 OLE, Week 20 OLE, Week 24 OLE, Week 28 OLE, Week 32 or 38 OLE (depending if entry was after extended induction phase), EoT up to 4 years (variable)
Population: FAS, separated by entry in OLE, data only shown if number of patients included in analysis ≥ 50 per visit
Measure: Median (Full Range); unit: mg/L
Arm/Group | 30 mg IMU-838 (Open-label Phase)
Number analyzed (Participants) | 190
mg/L
  Entry in OLE after (extended) induction phase - Baseline: number analyzed (Participants) | 115
  Entry in OLE after (extended) induction phase - Baseline | 5.20 [0.3 to 69.9]
  Entry in OLE after (extended) induction phase - Visit 1 (Week 4 OLE): number analyzed (Participants) | 101
  Entry in OLE after (extended) induction phase - Visit 1 (Week 4 OLE) | 3.30 [0.3 to 41.8]
  Entry in OLE after (extended) induction phase - Visit 2 (Week 8 OLE): number analyzed (Participants) | 89
  Entry in OLE after (extended) induction phase - Visit 2 (Week 8 OLE) | 2.30 [0.3 to 71.9]
  Entry in OLE after (extended) induction phase - Visit 3 (Week 12 OLE): number analyzed (Participants) | 83
  Entry in OLE after (extended) induction phase - Visit 3 (Week 12 OLE) | 2.40 [0.3 to 37.3]
  Entry in OLE after (extended) induction phase - Visit 4 (Week 16 OLE): number analyzed (Participants) | 77
  Entry in OLE after (extended) induction phase - Visit 4 (Week 16 OLE) | 2.60 [0.3 to 178.9]
  Entry in OLE after (extended) induction phase - Visit 5 (Week 20 OLE): number analyzed (Participants) | 68
  Entry in OLE after (extended) induction phase - Visit 5 (Week 20 OLE) | 3.60 [0.3 to 46.1]
  Entry in OLE after (extended) induction phase - Visit 6 (Week 24 OLE): number analyzed (Participants) | 58
  Entry in OLE after (extended) induction phase - Visit 6 (Week 24 OLE) | 3.40 [0.3 to 26.0]
  Entry in OLE after (extended) induction phase - Visit 7 (Week 28 OLE): number analyzed (Participants) | 55
  Entry in OLE after (extended) induction phase - Visit 7 (Week 28 OLE) | 2.80 [0.3 to 39.5]
  Entry in OLE after (extended) induction phase - Visit 8 (Week 32 or 38 OLE): number analyzed (Participants) | 51
  Entry in OLE after (extended) induction phase - Visit 8 (Week 32 or 38 OLE) | 2.20 [0.3 to 49.9]
  Entry in OLE after (extended) induction phase - end of treatment (up to 4 years, variable): number analyzed (Participants) | 74
  Entry in OLE after (extended) induction phase - end of treatment (up to 4 years, variable) | 2.45 [0.3 to 46.5]
  Entry in OLE after maintenance phase - Baseline: number analyzed (Participants) | 75
  Entry in OLE after maintenance phase - Baseline | 1.90 [0.3 to 56.0]
  Entry in OLE after maintenance phase - Visit 1 (Week 10 OLE): number analyzed (Participants) | 60
  Entry in OLE after maintenance phase - Visit 1 (Week 10 OLE) | 1.55 [0.3 to 79.8]
  Entry in OLE after maintenance phase - Visit 2 (Week 20 OLE): number analyzed (Participants) | 50
  Entry in OLE after maintenance phase - Visit 2 (Week 20 OLE) | 1.25 [0.3 to 16.3]

ADVERSE EVENTS:
Time Frame: Adverse events were collected during each study period: induction phase up to 22 weeks, maintenance phase up to 50 weeks, open-label phase up to 4 years
Groups:
- 30 mg IMU-838 (Induction Phase): Two 15 mg tablets once daily of IMU-838 for 10 to 22 weeks.
  IMU-838: IMU-838 tablet
- 45 mg IMU-838 (Induction Phase): Two 22.5 mg tablets once daily of IMU-838 for 10 to 22 weeks.
  IMU-838: IMU-838 tablet
- 10 mg IMU-838 (Maintenance Phase): Two 5 mg tablets once daily of IMU-838 for up to 50 weeks.
Arm/Group | 10 mg IMU-838 (Induction Phase) | 30 mg IMU-838 (Induction Phase) | 45 mg IMU-838 (Induction Phase) | Placebo (Induction Phase) | 10 mg IMU-838 (Maintenance Phase) | 30 mg IMU-838 (Maintenance Phase) | Placebo (Maintenance Phase) | 30 mg IMU-838 (Open-label Phase)
All-Cause Mortality (participants affected / at risk) | 0/67 | 0/67 | 0/66 | 0/63 | 0/45 | 0/40 | 0/27 | 0/190
Serious Adverse Events (participants affected / at risk) | 2/67 | 5/67 | 5/66 | 0/63 | 3/45 | 2/40 | 1/27 | 14/190
Other Adverse Events (participants affected / at risk) | 8/67 | 7/67 | 12/66 | 13/63 | 7/45 | 6/40 | 2/27 | 24/190
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 10 mg IMU-838 (Induction Phase) (N=67) | 30 mg IMU-838 (Induction Phase) (N=67) | 45 mg IMU-838 (Induction Phase) (N=66) | Placebo (Induction Phase) (N=63) | 10 mg IMU-838 (Maintenance Phase) (N=45) | 30 mg IMU-838 (Maintenance Phase) (N=40) | Placebo (Maintenance Phase) (N=27) | 30 mg IMU-838 (Open-label Phase) (N=190)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhea hemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proctitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Volvulus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abscess limb (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colon gangrene (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peritonitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skull fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 (0) | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal colic (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary sarcoidosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 10 mg IMU-838 (Induction Phase) (N=67) | 30 mg IMU-838 (Induction Phase) (N=67) | 45 mg IMU-838 (Induction Phase) (N=66) | Placebo (Induction Phase) (N=63) | 10 mg IMU-838 (Maintenance Phase) (N=45) | 30 mg IMU-838 (Maintenance Phase) (N=40) | Placebo (Maintenance Phase) (N=27) | 30 mg IMU-838 (Open-label Phase) (N=190)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 5 (5) | 3 (3) | 3 (3) | 1 (1) | 1 (1) | 2 (2) | 5 (6)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 2 (2) | 1 (1) | 2 (2) | 2 (2) | 5 (5) | 1 (1) | 0 (0) | 14 (14)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 3 (3)
Headache (Nervous system disorders) | 3 (3) | 1 (1) | 1 (1) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 5 (7)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 5 (7) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-14): https://cdn.clinicaltrials.gov/large-docs/62/NCT03341962/Prot_SAP_000.pdf